CLINICAL TRIAL: NCT03042871
Title: Dosing Strategy of Intravitreal Ranibizumab for Myopia Choroidal Neovascularization: a Single Center Randomized Prospective Study
Brief Title: Dosing Strategy of Intravitreal Ranibizumab for Pathological Myopia Choroidal Neovascularization
Acronym: SMILE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Zhongshan Ophthalmic Center, Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Xiaoyan Ding, Professor,PhD,MD, Zhongshan Ophthalmic Center, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2015002
Record Dates: First submitted 2016-08-21; First posted 2017-02-03 (Estimated); Last update posted 2019-03-11 (Actual); Status verified 2019-03

CONDITIONS: Choroidal Neovascularization
Keywords: PM-CNV ,Ranibizumab, Dosing Strategy
MeSH Terms: conditions — Choroidal Neovascularization

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A (Active Comparator): Group A included 30 patients treated with one 0.5mg intravitreal ranibizumab injection. All patients were followed monthly for 12 months with additional injections performed as needed.
  Interventions: Drug: 0.5mg intravitreal ranibizumab
- Group B (Active Comparator): Group B included 30 patients treated with three monthly 0.5mg intravitreal ranibizumab injections. All patients were followed monthly for 12 months with additional injections performed as needed.
  Interventions: Drug: 0.5mg intravitreal ranibizumab

INTERVENTIONS:
Drug: 0.5mg intravitreal ranibizumab — Patients received ranibizumab (0.5mg, Novartis AG, Basel, Switzerland) via a pars plana transcleral injection through 30-gauge needle at 3.5 to 4mm of inferotemporal limbus. Levofloxacin eye drops ( Cravit Eye Drops, Santen, Japan) was instilled 4 times a day in the study eye before the treatment at least 1 day. Povidone-iodine (5%, Luofushan Pharmaceutical Co., China) was applied to the conjunctiva bulbi and the fornices for at least 3 minutes before injection. Patients were instructed to continue the levofloxacin eye drops 4 times a day for 3 days
  Other Names: IVR 0.5mg

SUMMARY:
The purpose of this study is to compare the efficacy (times of injection, change of visual acuity and Cva/ I) and safety (macular visual function and choroidal thickness) of different dosing of ranibizumab intravitreal injection (1+PRN vs. 3+PRN) in treating with pathological myopia choroidal neovascularization (PM-CNV).

DETAILED DESCRIPTION:
PM is a common disease in east asia, while PM-CNV affect 5%-10% PM patients.PM-CNV has specific characteristics, including small dimensions and limited exudative manifestations comparing with age-related macular degeneration. However, treatment regimen and re-treatment criteria follow the PrONTO protocol. The question of the optimal dose and treatment regimen in myopic CNV management is still unresolved. There is no unequivocal evidence suggesting hat PRN treatment is more effective than a loading phase followed by an as-needed variable dosage regimen.

ELIGIBILITY:
Inclusion Criteria:

* older then 18 years old
* refractive error ≥ -6.0 diopters or axial length ≥ 26.0mm
* active CNV due to high myopic which is the only reason cause visual loss confirmed by fluorescein fundus angiography
* BCVA ≥ 24.0 and ≤73 letters at a starting distance of 4 meters using Early Treatment Diabetic Retinopathy Study visual acuity chart.

Exclusion Criteria:

* history of (a) stroke,(b) laser photocoagulation involved macular area in study eye, (c) intraocular treatment with corticosteroids or intraocular surgery or anti vascular endothelial growth factor or verteporfin photodynamic therapy within 6 months in study eye, or (d) hypersensitivity to ranibizumab or fluorescein
* presence of active infectious disease or confirmed intraocular pressure ≥ 21.0 mmHg
* pregnant or nursing women
* uncontrolled high blood pressure ≥ 150/90 mmHg or uncontrolled fasting blood glucose ≥ 7 mmol/L

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2015-04; Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Injection Number | 12 months
  Total IRV injection number
Best corrected visual acuity (BCVA) | Change from baseline to 12 months

SECONDARY OUTCOMES:
Retinal sensitivities on microperimetry | Baseline and monthly after enrollment from baseline up to 12 months
Electrical response densities in the foveal on multifocal electroretinogram | Baseline, 3 months, 6 months and 12 months after enrollment.
Alterations of optic coherence tomography angiography | Baseline, 3 months, 6 months and 12 months after enrollment.
Retinal thickness on optic coherence tomography | Baseline and monthly after enrollment up to 12 months.
Leakage in lesion on fluorescein fundus angiography | Baseline, 3 months, 6 months and 12 months after enrollment.
Fixation stability on microperimetry | Baseline and monthly after enrollment from baseline up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoyan Ding, PhD, Study Chair — ZZhongShan Ophthalmic Center, Sun Yat-sen University
Locations (1):
- ZhongShan Ophthalmic Center, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Van Newkirk MR. The Hong Kong vision study: a pilot assessment of visual impairment in adults. Trans Am Ophthalmol Soc. 1997;95:715-49. PMID 9440191
- [Background] Yoshida T, Ohno-Matsui K, Yasuzumi K, Kojima A, Shimada N, Futagami S, Tokoro T, Mochizuki M. Myopic choroidal neovascularization: a 10-year follow-up. Ophthalmology. 2003 Jul;110(7):1297-305. doi: 10.1016/S0161-6420(03)00461-5. PMID 12867382
- [Background] Wong TY, Foster PJ, Hee J, Ng TP, Tielsch JM, Chew SJ, Johnson GJ, Seah SK. Prevalence and risk factors for refractive errors in adult Chinese in Singapore. Invest Ophthalmol Vis Sci. 2000 Aug;41(9):2486-94. PMID 10937558
- [Background] Chan WM, Ohji M, Lai TY, Liu DT, Tano Y, Lam DS. Choroidal neovascularisation in pathological myopia: an update in management. Br J Ophthalmol. 2005 Nov;89(11):1522-8. doi: 10.1136/bjo.2005.074716. PMID 16234465
- [Background] Jones D, Luensmann D. The prevalence and impact of high myopia. Eye Contact Lens. 2012 May;38(3):188-96. doi: 10.1097/ICL.0b013e31824ccbc3. PMID 22495679
- [Background] Miller DG, Singerman LJ. Vision loss in younger patients: a review of choroidal neovascularization. Optom Vis Sci. 2006 May;83(5):316-25. doi: 10.1097/01.opx.0000216019.88256.eb. PMID 16699445
- [Background] Sun J, Zhou J, Zhao P, Lian J, Zhu H, Zhou Y, Sun Y, Wang Y, Zhao L, Wei Y, Wang L, Cun B, Ge S, Fan X. High prevalence of myopia and high myopia in 5060 Chinese university students in Shanghai. Invest Ophthalmol Vis Sci. 2012 Nov 1;53(12):7504-9. doi: 10.1167/iovs.11-8343. PMID 23060137
- [Background] Nagaoka N, Shimada N, Hayashi W, Hayashi K, Moriyama M, Yoshida T, Tokoro T, Ohno-Matsui K. Characteristics of periconus choroidal neovascularization in pathologic myopia. Am J Ophthalmol. 2011 Sep;152(3):420-427.e1. doi: 10.1016/j.ajo.2011.03.002. Epub 2011 Jun 22. PMID 21696698
- [Background] Verteporfin in Photodynamic Therapy Study Group. Photodynamic therapy of subfoveal choroidal neovascularization in pathologic myopia with verteporfin. 1-year results of a randomized clinical trial--VIP report no. 1. Ophthalmology. 2001 May;108(5):841-52. doi: 10.1016/s0161-6420(01)00544-9. PMID 11320011
- [Background] Blinder KJ, Blumenkranz MS, Bressler NM, Bressler SB, Donato G, Lewis H, Lim JI, Menchini U, Miller JW, Mones JM, Potter MJ, Pournaras C, Reaves A, Rosenfeld P, Schachat AP, Schmidt-Erfurth U, Sickenberg M, Singerman LJ, Slakter JS, Strong HA, Virgili G, Williams GA. Verteporfin therapy of subfoveal choroidal neovascularization in pathologic myopia: 2-year results of a randomized clinical trial--VIP report no. 3. Ophthalmology. 2003 Apr;110(4):667-73. doi: 10.1016/s0161-6420(02)01998-x. PMID 12689884
- [Background] Nguyen QD, Shah S, Tatlipinar S, Do DV, Anden EV, Campochiaro PA. Bevacizumab suppresses choroidal neovascularisation caused by pathological myopia. Br J Ophthalmol. 2005 Oct;89(10):1368-70. No abstract available. PMID 16170134
- [Background] Wolf S, Balciuniene VJ, Laganovska G, Menchini U, Ohno-Matsui K, Sharma T, Wong TY, Silva R, Pilz S, Gekkieva M; RADIANCE Study Group. RADIANCE: a randomized controlled study of ranibizumab in patients with choroidal neovascularization secondary to pathologic myopia. Ophthalmology. 2014 Mar;121(3):682-92.e2. doi: 10.1016/j.ophtha.2013.10.023. Epub 2013 Dec 8. PMID 24326106
- [Background] Grunwald JE, Daniel E, Huang J, Ying GS, Maguire MG, Toth CA, Jaffe GJ, Fine SL, Blodi B, Klein ML, Martin AA, Hagstrom SA, Martin DF; CATT Research Group. Risk of geographic atrophy in the comparison of age-related macular degeneration treatments trials. Ophthalmology. 2014 Jan;121(1):150-161. doi: 10.1016/j.ophtha.2013.08.015. Epub 2013 Sep 29. PMID 24084496
- [Background] Kung YH, Wu TT, Huang YH. One-year outcome of two different initial dosing regimens of intravitreal ranibizumab for myopic choroidal neovascularization. Acta Ophthalmol. 2014 Dec;92(8):e615-20. doi: 10.1111/aos.12457. Epub 2014 Jun 12. PMID 24924911